CLINICAL TRIAL: NCT02013245
Title: Phase I Double Blind, Randomized, Controlled, Dose-Escalation Study to Evaluate the Safety and Immunogenicity of MTBVAC in Comparison With BCG in Elispot TB(ESAT-6, CFP10, PPD)- and HIV- Negative Volunteers
Brief Title: Dose-Escalation Study to Evaluate the Safety and Immunogenicity of MTBVAC Vaccine in Comparison With BCG Vaccine.
Acronym: MTBVAC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biofabri, S.L (Industry)
Collaborators: Universidad de Zaragoza (Other); Centre Hospitalier Universitaire Vaudois (Other); TuBerculosis Vaccine Initiative (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MTBVAC-01
Record Dates: First submitted 2013-12-03; First posted 2013-12-17 (Estimated); Results first posted 2017-03-24 (Actual); Last update posted 2017-03-24 (Actual); Status verified 2017-02

CONDITIONS: Tuberculosis; Healthy
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MTBVAC group 1 (Experimental): Intervention: MTBVAC live vaccine (low dose 5 x 10E03 CFU/0.1mL)
  Interventions: Biological: MTBVAC live vaccine
- MTBVAC Group 2 (Experimental): Intervention: MTBVAC live vaccine (middle dose 5 x 10E04 CFU/0.1mL)
  Interventions: Biological: MTBVAC live vaccine
- MTBVAC Group 3 (Experimental): Intervention: MTBVAC live vaccine (high dose 5 x 10E05 CFU/0.1mL)
  Interventions: Biological: MTBVAC live vaccine
- BCG Control Group (Active Comparator): Intervention: Commercially available BCG live vaccine (dose 5 x 10E05 CFU/0.1mL)
  Interventions: Biological: Commercially available BCG live vaccine

INTERVENTIONS:
Biological: MTBVAC live vaccine — Live-attenuated Mycobacterium tuberculosis vaccine
  Arms: MTBVAC Group 2; MTBVAC Group 3; MTBVAC group 1
Biological: Commercially available BCG live vaccine — Live-attenuated Mycobacterium bovis vaccine
  Arms: BCG Control Group

SUMMARY:
The purpose of this study is to test the safety and immunogenicity of MTBVAC as a potential substitute for BCG vaccination. BCG vaccination has indeed demonstrated its major limitation in inducing protection against tuberculosis (TB). Novel vaccines are essential to fight against the current world epidemics in tuberculosis and resistance to anti-TB drugs.

DETAILED DESCRIPTION:
A randomized, double-blind, controlled Phase I study conducted at CHUV, Lausanne, Switzerland, to compare MTBVAC to licensed BCG in healthy, PPD-negative adult male and female volunteers. The study involves random allocation of up to 36 subjects (4 vaccine groups of 9 volunteers fulfilling the inclusion criteria) to MTBVAC (tested at three separate doses) or standard dose BCG (on a 3 verum : 1control basis) in a dose-escalation manner to one of three cohorts. Each cohort includes 9 subjects set to receive MTBVAC lowest dose 5x10E03, or MTBVAC intermediate dose 5x10E04, or high dose 5x10E05 colony forming units (CFU) in 0.1 mL and 3 subjects set to receive standard dose BCG (5x10E05 CFU in 0.1 mL). A single intradermal injection is given in the non-dominant arm of each volunteer starting with the lowest MTBVAC dose. Each MTBVAC vaccine dose is administered staggered by cohort, starting with the cohort with the lowest MTBVAC dose level. After at least 35 days of follow-up within each cohort a safety review and evaluation by Independent Data Safety Monitoring Board provides go/no-go for vaccination of the subsequent cohorts if no safety issues as defined by preset stopping rules.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the Investigator believes that they can and will comply with the requirements of the protocol
* Subjects who have no evidence of exposition to BCG as demonstrated by a ELISPOT PPD assay along with no history of BCG vaccination and no BCG scar
* A male or female between, and including, 18 and 45 years of age at the time of the vaccination.
* Written informed consent obtained from the subject prior to any study procedure.
* If the subject is female, she must be of non-childbearing potential, or if she is of childbearing potential, she must practice adequate contraception
* Clinically acceptable laboratory values for blood tests.
* Seronegative for human immunodeficiency virus 1 and -2 (HIV-1/2) antibodies, p24 antigen, hepatitis B surface antigen (HBsAg), and hepatitis C virus (HCV) antibodies.
* No evidence of pulmonary pathology as confirmed by chest X-ray.
* No history of extrapulmonary TB.
* No history of previous contact with M. tuberculosis (latent tuberculosis) as demonstrated by a negative ELISPOT Tb (ESAT-6, CFP10) assay.

Exclusion Criteria:

* History of allergic reactions (significant IgE-mediated events) or anaphylaxis to previous immunisations (any vaccine).
* History of allergic disease or reactions
* History of previous administration of experimental Mycobacterium tuberculosis vaccines.
* Use of any investigational or non-registered product (drug or vaccine) in another experimental protocol other than the study vaccines within 30 days preceding the vaccination, or planned use during the study period.
* Any chronic drug therapy to be continued during the study period.
* Chronic administration of immunosuppressors or other immune-modifying drugs.
* Administration of any immunoglobulins, any immunotherapy and/or any blood products within the three months preceding the vaccination, or planned administrations during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition (including HIV) based on medical history and physical examination.
* Any condition or history of any acute or chronic illness or medication which, in the opinion of the Investigator, may interfere with the evaluation of the study objectives.
* A family history of congenital or hereditary immunodeficiency.
* A stay of more than 2 months in a highly endemic area (e.g. Eastern Europe (Romania, Bulgaria) and low-income countries) within 6 months prior to the screening visit or travel of more than 2 months foreseen in an area of high endemicity after the enrolment into the study.
* History of any neurologic disorders or seizures.
* History of chronic alcohol consumption and/or drug abuse.
* Major congenital defects.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: François Spertini, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arbues A, Aguilo JI, Gonzalo-Asensio J, Marinova D, Uranga S, Puentes E, Fernandez C, Parra A, Cardona PJ, Vilaplana C, Ausina V, Williams A, Clark S, Malaga W, Guilhot C, Gicquel B, Martin C. Construction, characterization and preclinical evaluation of MTBVAC, the first live-attenuated M. tuberculosis-based vaccine to enter clinical trials. Vaccine. 2013 Oct 1;31(42):4867-73. doi: 10.1016/j.vaccine.2013.07.051. Epub 2013 Aug 17. PMID 23965219
- [Background] Verreck FA, Vervenne RA, Kondova I, van Kralingen KW, Remarque EJ, Braskamp G, van der Werff NM, Kersbergen A, Ottenhoff TH, Heidt PJ, Gilbert SC, Gicquel B, Hill AV, Martin C, McShane H, Thomas AW. MVA.85A boosting of BCG and an attenuated, phoP deficient M. tuberculosis vaccine both show protective efficacy against tuberculosis in rhesus macaques. PLoS One. 2009;4(4):e5264. doi: 10.1371/journal.pone.0005264. Epub 2009 Apr 15. PMID 19367339
- [Background] Gonzalo-Asensio J, Mostowy S, Harders-Westerveen J, Huygen K, Hernandez-Pando R, Thole J, Behr M, Gicquel B, Martin C. PhoP: a missing piece in the intricate puzzle of Mycobacterium tuberculosis virulence. PLoS One. 2008;3(10):e3496. doi: 10.1371/journal.pone.0003496. Epub 2008 Oct 23. PMID 18946503
- [Background] Martin C, Williams A, Hernandez-Pando R, Cardona PJ, Gormley E, Bordat Y, Soto CY, Clark SO, Hatch GJ, Aguilar D, Ausina V, Gicquel B. The live Mycobacterium tuberculosis phoP mutant strain is more attenuated than BCG and confers protective immunity against tuberculosis in mice and guinea pigs. Vaccine. 2006 Apr 24;24(17):3408-19. doi: 10.1016/j.vaccine.2006.03.017. PMID 16564606
- [Background] Perez E, Samper S, Bordas Y, Guilhot C, Gicquel B, Martin C. An essential role for phoP in Mycobacterium tuberculosis virulence. Mol Microbiol. 2001 Jul;41(1):179-87. doi: 10.1046/j.1365-2958.2001.02500.x. PMID 11454210
- [Result] Spertini F, Audran R, Chakour R, Karoui O, Steiner-Monard V, Thierry AC, Mayor CE, Rettby N, Jaton K, Vallotton L, Lazor-Blanchet C, Doce J, Puentes E, Marinova D, Aguilo N, Martin C. Safety of human immunisation with a live-attenuated Mycobacterium tuberculosis vaccine: a randomised, double-blind, controlled phase I trial. Lancet Respir Med. 2015 Dec;3(12):953-62. doi: 10.1016/S2213-2600(15)00435-X. Epub 2015 Nov 17. PMID 26598141

RESULTS

PARTICIPANT FLOW:
Groups:
- MTBVAC Group 1: Intervention: MTBVAC live vaccine (low dose 5 x 10^3 CFU)
- MTBVAC Group 2: Intervention: MTBVAC live vaccine (middle dose 5 x 10^4 CFU)
- MTBVAC Group 3: Intervention: MTBVAC live vaccine (high dose 5 x 10^5 CFU)
- BCG Control Group: Intervention: Commercially available BCG live vaccine (dose 5 x 10^5 CFU)
Period: Overall Study
Arm/Group | MTBVAC Group 1 | MTBVAC Group 2 | MTBVAC Group 3 | BCG Control Group
Started | 9 | 9 | 9 | 9
Completed | 9 | 8 | 9 | 9
Not Completed | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: MTBVAC low dose group (5 x 10^3 CFU MTBVAC)
- Group 2: MTBVAC intermediate dose group (5 x 10^4 CFU MTBVAC)
- Group 3: MTBVAC high dose group (5 x 10^5 CFU MTBVAC)
- BCG Control Group: BCG standard dose group (5 x 10^5 CFU BCG)
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | BCG Control Group | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 9 | 9 | 36
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (9.6) | 28.2 (3.2) | 27.1 (6.1) | 25.6 (3.4) | 27.2 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 7 | 6 | 22
  Male | 6 | 3 | 2 | 3 | 14
Region of Enrollment [Number; unit: participants]
  Switzerland | 9 | 9 | 9 | 9 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events up to 210 Days After Vaccination
Description: Safety and reactogenicity for all subjects as determined by:
  * Occurrence of solicited symptoms during the 7-day follow-up period following vaccination and occurrence of unsolicited symptoms during the 210-day follow-up period following vaccination.
  * Occurrence of grade 3 vaccine related local and general symptoms during the 210-day follow-up period following vaccination and occurrence of serious adverse events throughout the entire study period.
  * Haematological and biochemical safety test levels prior and after vaccination
Time Frame: 7 months follow up
Measure: Number; unit: participants
Groups:
- BCG Control Group: Intervention: Commercially available BCg live vaccine (standard dose 5 x 10^5 CFU)
Arm/Group | MTBVAC Group 1 | MTBVAC Group 2 | MTBVAC Group 3 | BCG Control Group
Number analyzed (Participants) | 9 | 9 | 9 | 9
participants | 9 | 9 | 9 | 9

2. Secondary Outcome: Number of Participants With Three-cytokine-positive CD4+ T-cell Response
Description: Measure of the kinetics of CD4+ T-cell responses to MTBVAC or BCG vaccination by tracking the expression of IFNγ, TNFα and IL-2 upon stimulation with live MTBVAC or BCG
Time Frame: Day 28
Population: Number of Participants with Three-cytokine-positive CD4+ T-cell Response (per protocol analysis)
Measure: Number; unit: participants
Arm/Group | MTBVAC Group 1 | MTBVAC Group 2 | MTBVAC Group 3 | BCG Control Group
Number analyzed (Participants) | 9 | 8 | 9 | 9
participants | 0 | 0 | 4 | 1

ADVERSE EVENTS:
Time Frame: Solicited local and systemic adverse events: within 7 days of vaccination (diary card). Unsolicited local and systemic adverse events at days 0, 7, 28, 56, 90, 150 and 210
Description: Safety was assessed based on a collection of solicited local (injection site pain, erythema, induration, pruritus and discharges) and systemic (fever, headache, fatigue, musculoskeletal pains, gastrointestinal symptoms) adverse events (AEs) within 7 days of vaccination (diary card). Unsolicited local and systemic AEs as well as serious AEs (SAEs) were collected during the entire study period.
Arm/Group | MTBVAC Group 1 | MTBVAC Group 2 | MTBVAC Group 3 | BCG Control Group
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 9/9 | 9/9 | 9/9 | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MTBVAC Group 1 (N=9) | MTBVAC Group 2 (N=9) | MTBVAC Group 3 (N=9) | BCG Control Group (N=9)
Pain at injection site (Skin and subcutaneous tissue disorders) | 3 | 5 | 5 | 8 — Pain at injection site
Erythema (Skin and subcutaneous tissue disorders) | 5 | 8 | 8 | 7 — Erythema at injection site
Induration (Skin and subcutaneous tissue disorders) | 5 | 7 | 8 | 9 — Induration at injection site
Pruritis (Skin and subcutaneous tissue disorders) | 3 | 3 | 1 | 2 — Pruritis at site of injection
Discharge (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 4 — Discharge from site of injection
Headache (General disorders) | 5 | 4 | 3 | 3 — General headache related or unrelated to vaccination
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 5 | 2 | 5 | 2 — Musculoskeletal pain
Fatigue (General disorders) | 7 | 4 | 3 | 4
Digestive (Gastrointestinal disorders) | 1 | 3 | 2 | 3
Fever (General disorders) | 1 | 4 | 3 | 1

LIMITATIONS AND CAVEATS:
This is a first-in-human Phase 1 trial designed to evaluate the safety and tolerability profile of MTBVAC in comparison to BCG.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less